CLINICAL TRIAL: NCT04764500
Title: Developing Microbials to Fight Extended-spectrum Beta-lactamase (ESBL)-Producing Escherichia Coli
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Gebert Rüf-Stiftung (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019-00044; am21Egli
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Extended Spectrum Beta Lactamases (ESBL) E. Coli
Keywords: Antibiotic resistance; pan-sensitive strains (non-ESBL E. coli); multidrug resistant E. coli strains; ESBL E. coli displacement; multidrug resistant Enterobacteriaceae
MeSH Terms: conditions — Escherichia coli Infections | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bacterial isolates and -80°C stool samples. Serum samples and blood cells may be used for antibody analysis and blood cell analysis (incl. B-cell immortalization for monoclonal antibody generation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- travellers to Southeast Asia: Clients planning to travel to Southeast Asia will be recruited
  Interventions: Other: examination of stool sample; Other: patient questionnaire; Other: examination of blood sample

INTERVENTIONS:
Other: examination of stool sample — Each participant provides stool samples before and after travelling, after 2, 4, 6, 8, 10, 12, 16, 20 and 52 weeks. Stool samples will be used for isolating both a) ESBL E. coli strains and b) pan-sensitive E. coli strains. Part of the stool sample is stored for isolation of further E. coli clones and microbiota analysis of the isolation of other microbiota strains. All found Enterobacteriaceae will be screened for additional resistance such as Carbapenem and Colistin. In case of a specific resistance, this will be confirmed with additional phenotypic and genotypic tests such as ROSCO disk and polymerase chain reaction (PCR) based panel and whole genome sequencing in order to detect specific resistance mechanisms and genes. Bacteria will be sequenced using Illumina and Nanopore based sequencing. Bioinformatic analysis will allow to determine the whole bacterial genome with containing resistance genes and also describe the microbiota diversity over time in single individuals.
Other: patient questionnaire — Each participant will have to provide a questionnaire before and after travelling, as well after 2, 4, 6, 8, 10, 12, 16, 20 and 52 weeks.
Other: examination of blood sample — Each participant will have to provide a blood sample before and after travelling and after 6, 12 and 20 weeks. A serum sample (5mL) for antibody measurement and a 50 ml blood sample for recovery of peripheral blood mononuclear cells (PBMCs in 6 CPTs) for cell mediated immunity will be collected. Serum and PBMCs will allow the analysis of anti-E. coli humoral and cellular responses in order to characterize the individual immune response to specific bacteria over time. Single nucleotide polymorphisms associated with humoral and cellular immune responses will be characterized and linked to immunological and clinical phenotypes and endpoints of the study.

SUMMARY:
This study is to identify and isolate well-defined microbials (non-ESBL E. coli) in an observational setting exploring natural gastrointestinal decolonization of humans colonized with ESBL E. coli.

DETAILED DESCRIPTION:
Antibiotic resistance is a severe threat to contemporary medicine. Effective approaches to fight multi-drug resistant pathogenic bacteria are needed.

This clinical observational study is to investigate whether express extended spectrum beta lactamases (ESBL) E. coli colonizing the human gut can be out-competed by other, ideally pan-sensitive strains (non-ESBL E. coli).

ELIGIBILITY:
Inclusion Criteria:

* travelling to Southeast Asia (India, Bhutan, Nepal, Bangladesh, Myanmar, Thailand, Laos, Cambodia, Vietnam) for a maximum of 4 weeks.

Exclusion Criteria:

* other travelling destinations than mentioned above
* antibiotic use at the first sampling time
* Participants who are not colonized will serve as a control group for microbiome comparison

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clients planning to travel to Southeast Asia will be recruited while receiving pre-travel health advice at the travel clinic of the Swiss Tropical and Public Health Institute in Basel.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
proportion of patients being "naturally" decolonized from ESBL E. coli | 18 months
  proportion of patients being "naturally" decolonized from ESBL E. coli at the end of the study period at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Egli, PD Dr. med., Principal Investigator — Division of Clinical Microbiology, University Hospital Basel
Locations (1):
- University Hospital Basel, Division of Clinical Microbiology, Basel, Switzerland